CLINICAL TRIAL: NCT01398904
Title: Attentional Bias in Body Dysmorphic Disorder
Acronym: VAB
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sabine Wilhelm, Director, OCD & Related Disorders Program, Massachusetts General Hospital
Other Study IDs: 2010P002912
Record Dates: First submitted 2011-07-15; First posted 2011-07-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Body Dysmorphic Disorders
Keywords: BDD
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Body dysmorphic disorder (BDD) Participants: Participants must be 18 years or older with a primary diagnosis of body dysmorphic disorder (BDD), a BDD Yale-Brown Obsessive Compulsive Scale (BDDY-BOCS) score of >20, and a primary facial/head concern. Participants must have the ability to provide informed consent and understand study staff.
- Healthy Controls: Males and females 18 years of age or older with ability to provide informed consent and understand study staff.

SUMMARY:
Body Dysmorphic Disorder (BDD) participants will demonstrate greater attentional biases as compared to healthy control (HC) participants. Greater attention bias will be associated with greater distress. Greater attention bias will be associated with greater symptom severity.

ELIGIBILITY:
Inclusion Criteria for BDD and healthy control participants:

* males and females 18 years of age or older
* sufficient fluency of English to understand study staff, procedures, and questionnaires
* ability to provide informed consent

Inclusion for BDD participants only;

* primary diagnosis of Diagnostic and Statistical Manual 4th Edition (DSM-IV-TR) BDD
* BDD Yale-Brown Obsessive Compulsive Disorder score (Y-BOCS) of > 20
* primary facial/head concern

Exclusion Criteria:

* Major medical or neurological conditions
* schizophrenia, schizoaffective disorder, or any other current lifetime DSM-IV psychotic disorder that is not attributable to delusional BDD
* current suicidality
* current homicidality

Exclusion criteria for healthy controls:

* Any current Axis I psychiatric illness
* history of BDD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 40 participants, consisting of 20 BDD participants and 20 matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Attention Pattern | Day 2
  Gaze tracking via an Eyelink II eye tracker will determine perception of visual information.

SECONDARY OUTCOMES:
Subjective Units of Distress Scale (SUDS) | Day 2
  Participants will provide a distress score based on the facial images observed.
Facial Attractiveness | Day 2
  Using a 9-point Likert scale, participants will rate the perceived most attractive and unattractive feature of their own and the control face.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, Ph. D., Principal Investigator — Massachusetts General Hospital; Jennifer Greenberg, Psy. D., Study Director — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Deckersbach T, Savage CR, Phillips KA, Wilhelm S, Buhlmann U, Rauch SL, Baer L, Jenike MA. Characteristics of memory dysfunction in body dysmorphic disorder. J Int Neuropsychol Soc. 2000 Sep;6(6):673-81. doi: 10.1017/s1355617700666055. PMID 11011514
- [Background] Phillips KA. Quality of life for patients with body dysmorphic disorder. J Nerv Ment Dis. 2000 Mar;188(3):170-5. doi: 10.1097/00005053-200003000-00007. PMID 10749282
- [Background] Phillips KA, Coles ME, Menard W, Yen S, Fay C, Weisberg RB. Suicidal ideation and suicide attempts in body dysmorphic disorder. J Clin Psychiatry. 2005 Jun;66(6):717-25. doi: 10.4088/jcp.v66n0607. PMID 15960564
- [Background] Phillips KA, Menard W, Fay C, Pagano ME. Psychosocial functioning and quality of life in body dysmorphic disorder. Compr Psychiatry. 2005 Jul-Aug;46(4):254-60. doi: 10.1016/j.comppsych.2004.10.004. PMID 16175755
- [Background] Savage CR, Baer L, Keuthen NJ, Brown HD, Rauch SL, Jenike MA. Organizational strategies mediate nonverbal memory impairment in obsessive-compulsive disorder. Biol Psychiatry. 1999 Apr 1;45(7):905-16. doi: 10.1016/s0006-3223(98)00278-9. PMID 10202579
- [Background] Kelly MM, Walters C, Phillips KA. Social anxiety and its relationship to functional impairment in body dysmorphic disorder. Behav Ther. 2010 Jun;41(2):143-53. doi: 10.1016/j.beth.2009.01.005. Epub 2009 Oct 7. PMID 20412881
- [Background] Maner JK, Holm-Denoma JM, Van Orden KA, Gailliot MT, Gordon KH, Joiner TE Jr. Evidence for attentional bias in women exhibiting bulimotypic symptoms. Int J Eat Disord. 2006 Jan;39(1):55-61. doi: 10.1002/eat.20222. PMID 16231350
- [Background] Roefs A, Jansen A, Moresi S, Willems P, van Grootel S, van der Borgh A. Looking good. BMI, attractiveness bias and visual attention. Appetite. 2008 Nov;51(3):552-5. doi: 10.1016/j.appet.2008.04.008. Epub 2008 Apr 15. PMID 18495295
- [Background] Carey P, Seedat S, Warwick J, van Heerden B, Stein DJ. SPECT imaging of body dysmorphic disorder. J Neuropsychiatry Clin Neurosci. 2004 Summer;16(3):357-9. doi: 10.1176/jnp.16.3.357. PMID 15377744
- [Background] Janelle CM, Hausenblas HA, Fallon EA, Gardner RE. A visual search examination of attentional biases among individuals with high and low drive for thinness. Eat Weight Disord. 2003 Jun;8(2):138-44. doi: 10.1007/BF03325003. PMID 12880191